CLINICAL TRIAL: NCT00516022
Title: Mistletoe as Complementary Treatment in Patients With Advanced Non-small-cell Lung Cancer (NSCLC), Treated With Carboplatin/Gemcitabine Chemotherapy Combination: Randomized Phase II Study
Brief Title: Mistletoe as Complementary Treatment in Patients With Advanced Non-small-cell Lung Cancer (NSCLC), Treated With Carboplatin/Gemcitabine Chemotherapy Combination.
Acronym: Iscador
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Weleda AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mistletoe.ctil
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigator product (Experimental): The patients randomized to this arm will receive the IP injections at home 3 times a week (the patients will inject the IP themselves).
  Interventions: Drug: Mistletoe extract
- Control (Other): The patients randomized to this arm will continue to receive chemotherapy as usual without further treatment (unless prescribed by the Doctor).
  Interventions: Drug: Mistletoe extract

INTERVENTIONS:
Drug: Mistletoe extract — The drug will be administered 3 times a week at home.
  Other Names: There's no drug to be administered in the control group.

SUMMARY:
Mistletoe extract is one of the most common complementary treatments used in Europe. Recent basic studies reported tumor response and survival prolongation in number of treatments with Mistletoe preparations. There are evidence based data for using this drug as side effect reducer when use in combination with chemotherapy regimen treatment. Other clinical data, although not well based is that complementary treatment when used in combination with the common oncology treatment has tumor response effect. Combinations with platinum compound and a third generation cytotoxic agent have been accepted as 'standard of care' for patients with advanced NSCLC. The combination of platinum compound and one of the new agents are associated with response rates of 30-40% and a median survival of 8-11 months for advanced NSCLC patients with good performance status.

Study objective: Improvement in QOL, Improvement in the toxicity profile of the chemotherapy treatment.

DETAILED DESCRIPTION:
The study design is to include 90 subjects. All subjects are treated with the common chemotherapy treatment. 50 percent will be treated with Iscador as combination with their common chemotherapy regimen. Common chemotherapy regimen used for NSCLC: Carboplatin and Gemcitabine. All study participants will receive this same chemotherapy regimen. This chemotherapy treatment is given every 3 weeks for up to 6 treatment cycles. The first day of the first treatment cycle, the combination of both Carboplatin and Gemcitabine will be administered. After a week (day 8 of treatment cycle) only Gemcitabine will be administered. Drugs would be calculated according to patient's body mass, renal function and general appearance. Once the patient signed Informed Consent he is assigned randomly to be treated with/without the injections of Mistletoe (called "Iscador"). Patient will receive the study medication (Iscador) as an intravenous injection that can be self injected or injected by any other of the family. Injections would be administered with low dose at the first week of the first treatment cycle and then, dose would be escalated, so as to check high sensitivity to the drug. Dosage would include: 2 injections of 0.1 mg, 2 injections of 0.1 mg and 2 injections of 1 mg. After that, treatment would continue with dosage of 10 g once every 2 days.

Patients from both treatment arms would be asked to fill-out QOL questionnaires at every treatment cycle and at follow-up visit after.

Study Primary Objectives:

1. Improvement in QOL
2. Improvement in the toxicity profile of the chemotherapy treatment

Secondary Objectives:

1. Improvement in time to tumor progression (TTP) and survival.
2. Safety profile of mistletoe extract with combination of chemotherapy treatment

This is a single center study, randomized phase II, with patients with advanced NSCLC treated with carboplatin/gemcitabine chemotherapy combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Histology proven of NSCLC
3. Stage IIIB or IV (TNM classification)
4. Performance status < 2 (ECOG classification
5. Measurable disease with one or more disease sites measured by computed tomography (CT)
6. Life expectancy of more than 12 weeks.
7. Treatment combination of gemcitabine/carboplatin (GC)
8. Sign of written informed consent -

Exclusion Criteria:

1. Prior chemotherapy
2. Prior radiation- allowed as long as the treatment was not targeted only site of measurable disease and given more than 3 weeks before entry the trial.
3. Central nervous system metastases
4. Hypercalcemia
5. Other life threatening medical conditions
6. Patients not able to comply with s.c. injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Quality Of Life | During the trial
  To check the effect of the treatment(or lack of it) on the quality of life of the patients enrolled to the trial.
Improvement in QOL. Improvement in the toxicity profile of the chemotherapy treatment | During all the trial
  To check on the difference in QoL of all patients.

SECONDARY OUTCOMES:
Objective Response | During all the duration of the trial
  The patients are asked to answer questions and the doctor will check blood works resolts.
Improvement in time to tumor progression (TTP) and survival Safety profile of mistletoe extract with combination of chemotherapy treatment | During duration of all the trial
  Looking out for difference in toxicity profile of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Gil Bar-Sela, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel